CLINICAL TRIAL: NCT02412007
Title: A Prospective Study (RCT) to Evaluate the Efficacy of an Individualized Comprehensive Home-Centred Activity Based Therapy for Children With Diplegic Cerebral Palsy
Brief Title: Individualized Comprehensive Home-Centred Activity Based Therapy for Children With Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, DR J N GOSWAMI, Senior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Activity Based Therapy in CP
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Diplegic Cerebral Palsy
Keywords: spastic diplegia;cerebral palsy;activity based therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Individualized comprehensive home centred activity based programme. Simple activities would be advised on the basis of child's individual characteristics and parental expectations. These would include but would not be limited to (a) Standing up from squatting position to catch an object of interest.
  (b) Squatting from standing position to pick an object of interest. (c) Walking to reach an object of interest. (d) Climbing up steps to get an object of interest. (e) Climbing down steps to keep the above object of interest. (f) Cycling (g) Kicking a football (h) Dancing
  Interventions: Other: Individualized comprehensive home centred activity based programme
- Group B (Active Comparator): Conventional Physiotherapy Conventional physiotherapy would include and would not be limited to
  1. Passive stretching exercises for spasticity reduction
  2. Gait exercises
  3. Walking on treadmill
  4. Lower limb strengthening exercises
  5. Exercises for balance improvenet
  Interventions: Other: Individualized comprehensive home centred activity based programme

INTERVENTIONS:
Other: Individualized comprehensive home centred activity based programme — Simple activities would be advised on the basis of child's individual characteristics and parental expectations. These would include but would not be limited to
  1. Standing up from squatting position to catch an object of interest.
  2. Squatting from standing position to pick an object of interest.
  3. Walking to reach an object of interest.
  4. Climbing up steps to get an object of interest.
  5. Climbing down steps to keep the above object of interest.
  6. Cycling
  7. Kicking a football
  8. Dancing
  Other Names: Activity Based Therapy

SUMMARY:
Activity based therapy is gaining interest for rehabilitation of children with cerebral palsy (CP). A home-based comprehensive programme structured on the principles of activity based therapy seems to hold promise in the field of rehabilitation of children with diplegic CP.This may reduce morbidity as well as promote better quality of life in these children . In this backdrop our study has been planned with an aim to evaluate the efficacy of a comprehensive home-centred activity based programme for children with diplegic CP.

DETAILED DESCRIPTION:
Study settings:

This study will be conducted on children enrolled in the Outpatient Clinic of Department of Pediatrics, Post Graduate Institute of Medical Education and Research, Chandigarh and the associated Outpatient Department of PRAYAAS (A project of Indian Council for Child Welfare) located at Dakshin Marg, Sector 38 B, Chandigarh which is a rehabilitation centre for children with cerebral palsy where the neurology unit of the department provides outreach services.

Study Period:

Oct 2014 to Dec 2015

Study population:

Consecutive children between 5 to 12 yrs age diagnosed as spastic diplegic cerebral palsy (as per the standard definition) brought to Outpatient Clinic of Department of Pediatrics, Post Graduate Institute of Medical Education and Research, Chandigarh and the associated Outpatient Department of PRAYAAS located at Dakshin Marg, Sector 38 B, Chandigarh.

Sample Size:

Keeping α=0.05.Power=80% Assumption: The intervention will result in 60metres change in distance covered.

S.D. from previous study for (Gross Motor Function Classification System)GMFCS II =77 Hence, we would need 27 children in each group. Assuming a loss of follow-up of 5 patients, targeted sample size is 59.Therefore we would require 30 patients per group .

Study design:

Endpoint: Efficacy, Feasibility Intervention model: Parallel group assignment Primary Purpose: Physiotherapy Masking: Intervention - Open label Outcome assessment- Blinded Assessment of Data- Blinded

Eligibility All children aged 5 to 12 years diagnosed with spastic diplegic cerebral palsy will be eligible for enrolment in the study. For the study, spastic diplegia would include those who have bilateral motor impairment affecting both lower extremities more than the upper extremities with objective clinical signs of both hyperreflexia and spasticity.

Primary Outcome variables At six months Change in distance covered as measured by 6 minute walk test (in metres)

Secondary Outcome variables:

At three months and six months

1. Change in Modified Ashworth Scale Scores
2. Change in Modified Tardieu Scale Scores
3. Change in 10metre fast walk score (in seconds)
4. Change in GMFM D & E Scores.
5. Change in Cerebral Palsy Quality of Life(CPQoL) (Primary Caregiver) Scores At three months Change in distance covered as measured by 6 minute walk test (in metres)

Methodology:

Patient flow Consecutive children of both sexes between 5-12 years with a clinical diagnosis of spastic cerebral palsy will be examined by the investigator and those meeting the inclusion criteria would be enrolled in the study.An informed consent would be taken from the parents or guardian prior to enrollment in the study. Clinical and demographic data will be recorded on a structured Performa for each child including age, sex, weight, detailed antenatal and birth history, complications during prenatal and neonatal period, detailed developmental history, and family history of any neurological conditions and presence of any known comorbidity of cerebral palsy.

Randomization Children would be randomized into two groups by using randomization table. They would be classified into either Group A or Group B Intervention Group A Children included in Group A would be advised to carry out an individualized comprehensive home centred activity based programme. The investigator would interact with the primary care-giver and record the parent's anticipated goals in terms of the child's lower limb functioning; specifically gait, spasticity and daily functioning. The child would be clinically examined thoroughly to see for impairments. Subsequently a comprehensive individualized activity based programme will be decided upon by discussion between the investigator, physiotherapist and occupational therapist and primary care-giver so that it is acceptable and feasible to be performed at home in a resource limited setting.

The programme would include simple activities which would be advised on the basis of child's individual characteristics and parental expectations. These would include but would not be limited to

1. Standing up from squatting position to catch an object of interest.
2. Squatting from standing position to pick an object of interest.
3. Walking to reach an object of interest.
4. Climbing up steps to get an object of interest.
5. Climbing down steps to keep the above object of interest.
6. Cycling
7. Kicking a football
8. Dancing

The total duration of activity would be one hour to start with and could be repeated to three times a day.

The frequency of activity would be at least five days a week . Parents would be advised that in case the child has any acute illness, fever, muscle pain, they should withhold the sessions and seek early medical consultation at PGIMER or contact the investigator for advice.

Group B Children included in Group B would continue to receive rehabilitative measures that they already are on in the form of conventional physiotherapy which would include and would not be limited to

1. Passive stretching exercises for spasticity reduction
2. Gait exercises
3. Walking on treadmill
4. Lower limb strengthening exercises
5. Exercises for balance improvement No extra intervention would be advised to this group as a part of the study. At the completion of the study, if comprehensive individualized home-centred activity based therapy is found to be efficacious, the same will be offered to children classified under Group B .

Follow-up Schedule

All children would be followed at set intervals from initiation of therapy as noted below:

1. Two weeks (telephonic/home visit)
2. Three months : Physical follow-up
3. Six months: Physical follow-up The first visit would be primarily aimed at reinforcing the techniques of therapy and clarifying parent's doubts.

Compliance would be assessed by reviewing written log of activity done at home.

At three-month visit the children would be clinically examined and following records made:

(a) 6 minute walk score (in metres) (b) Modified Ashworth Score (b) Modified Tardieu Score (c) 10metre fast walk score (in metres) (d) GMFM D Score (e) GMFM E Score (f) CPQoL (Primary Care giver) Score

At six-month visit the children would be clinically examined and following records made:

1. Modified Ashworth Score
2. Modified Tardieu Score
3. 10metre fast walk score (in metres)
4. GMFM D Score
5. GMFM E Score
6. CPQoL(Primary Caregiver) Score

Statistical Analysis

Statistics: Data record would be done in a Microsoft Excel spreadsheet (Microsoft Office, Microsoft Corp., Seattle, WA, USA).

(i) Descriptive: Mean/Median/Range/Standard Deviation/Frequencies would be used to describe the demographic profile of patients and their comorbidities.

(iii) Comparative: Appropriate tests would be employed

Ethical justification The study consists of a comparative analysis between the effects of conventional physiotherapy and those of a comprehensive individualized home-centred activity-based programme on children with spastic diplegia. All children would be examined in detail and either of the interventions would be advised after random selection. Both of these interventions are beneficial and hence every child enrolled would be benefited. The children would be evaluated for co-morbidities and appropriate therapy advised as and when needed. This study would be beneficial in the long term in designing and recommending an effective exercise programme for spastic diplegics.

No additional investigations will be done for the purpose of the study. Parents will have the privilege to withdraw their child from the study at any point of study period. This will in no way affect the standard protocol of management of the child. Children enrolled in the study would benefit by undergoing a comprehensive and standardized evaluation of their disabilities and getting the benefits of a regular rehabilitative programme.

ELIGIBILITY:
Inclusion Criteria:

1. Children of either sex aged 5 to 12 years clinically diagnosed to have spastic diplegic cerebral palsy .
2. GMFCS either II or III
3. Minimum visual acuity of 6/60
4. Ability to follow simple single step commands
5. Either parent should be willing and capable of following instructions and maintaining activity log.

Exclusion Criteria:

1. Children with fixed contractures and deformities in lower limbs affecting stance and gait.
2. Children who have received botulinum toxin injection or undergone orthopaedic corrective surgery in the past one year.
3. Children with concomitant chronic systemic illnesses that can interfere with execution of physiotherapy or activity based therapy.
4. Children with any acute illness.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in distance covered as measured by 6 minute walk test (in metres) | six months
  The test is performed on a quadrangular ,plain floor which has a marked rectangular area,the perimeter of which is thirty four metres.Subject and his/her attendant is initially given demonstration and then he/she is made to walk along the marked surface continuously for six minutes and the same is videographed..The distance covered is measured and recorded.

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale Score | 3 months; 6 months
Change in Modified tardieu Scale Score | 3 months; 6 months
Change in 10metres fast walk score | baseline, 3 months; 6 months
  Child is made to walk 10 metres on a plain marked surface and the time taken for the same is recorded.The same is videographed.This is done at enrollment and 3 months and 6 months after enrolment
Change in Gross Motor Function Measure 88 D & E Scores (GMFM-88 D & E) | 3 months; 6 months
Change in Cerebral Palsy Quality of Life (Primary Care Giver ) Score (CPQoL) | 3 months; 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof Pratibha Singhi, MD, Study Director — Post Graduate Institute of Medical Education and Research,Chandigarh,India
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India